CLINICAL TRIAL: NCT04048863
Title: Assessment of the Effect of B. Braun Peripheral Advantage Program on Complications, Indwell Time and First Stick Success of PIVC Therapy
Brief Title: Effect of B. Braun Peripheral Advantage Program on Complications, Indwell Time and First Stick Success of PIVC Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated due to recruitment futility resulting from the significant impact of the COVID-19 pandemic to our intended study population and facility personnel.
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: US-N-H-1801
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Complications Associated With Device

STUDY DESIGN:
Intervention Model Description: The study will be divided into 4 Stages: 3 Clinical Stages and 1 Educational Stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Stage 1 Baseline (Active Comparator): Study site to use standard of care PIVC device(s) and procedure(s) on patients.
  Interventions: Device: Hospital Standard of Care
- Stage 2 Education (Other): RN education and training in the use of B. Braun PIVC products, devices and procedures.
  Interventions: Device: B. Braun Peripheral Advantage (PA) Program
- Stage 3 Run-In (Other): Familiarization of study RNs with the B. Braun devices and procedures in a clinical setting.
  Interventions: Device: B. Braun Peripheral Advantage (PA) Program
- Stage 4 Post-Education (Other): Study site uses B. Braun PIVC device(s) and procedure(s) on patients.
  Interventions: Device: B. Braun Peripheral Advantage (PA) Program

INTERVENTIONS:
Device: B. Braun Peripheral Advantage (PA) Program — B. Braun PA includes: Christie VeinViewer® Vision2 , Introcan Safety® IV Catheters, STEADYCare™ Smallbore Extension Set, and the PA Education
  Arms: Stage 2 Education; Stage 3 Run-In; Stage 4 Post-Education
Device: Hospital Standard of Care — Standard of Care for PIVC access per hospital protocol
  Arms: Stage 1 Baseline

SUMMARY:
Single sequence clinical study designed to evaluate the effectiveness of B. Braun PA on improved clinical outcomes, indwell time and first stick success of PIVC using B. Braun Peripheral Advantage (PA) by Registered Nurses (RNs).

The study will be conducted in the Emergency Department (ED) and/or Medical Surgical (MS) floor(s)/unit(s) in multiple hospitals.

ELIGIBILITY:
Inclusion Criteria:

* RNs must complete all of the required B. Braun trainings in Stage 2 in order to participate in Stages 3 and 4.

Subjects must meet all of the following Inclusion Criteria:

1. Male or female aged ≥18 years;
2. The subject or the subject's LAR voluntarily agrees that the subject will participate in this study and is able to understand and sign the Informed Consent Form (ICF);
3. Have a medical condition that requires a PIVC anticipated to last for at least 48 hours;
4. Have intact skin at the site of insertion;
5. If the patient has an existing IV in one arm he/she must have a viable contralateral arm for additional PIVC insertion.

Exclusion Criteria:

Subjects must not meet any of the following Exclusion Criteria:

1. Are currently participating in another medical device or pharmaceutical study;
2. In the opinion of the Investigator, would not be suitable candidates for this study;
3. The subject or his/her LAR is an employee of the Investigator or study center, or the sponsor, or have direct involvement in the study or other studies under the direction of that Investigator or study center, or are a family member of the employees or the Investigator;
4. Have a laboratory confirmed bloodstream infection within 48 hours prior to participation in the study. The assessment is based on clinical observations and not routine for all subjects;
5. Patient has an existing non study related IV;
6. Was removed from any Stage of the study due to an AE associated with the PIVC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla M Jaekel, RN, Principal Investigator — Mayo Clinic - La Crosse, WI
Locations (1):
- Mayo Clinic, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated during Stage 1 for recruitment futility. Stages 2 through 4 were not conducted.
  44 subjects (patients) were consented in Stage 1, however one subject failed inclusion/exclusion criteria. Thus 43 subjects received study procedures.
Groups:
- Stage 1 Baseline: Study site to use standard of care PIVC device(s) and procedure(s) on patients.
  For this study, PARTICIPANTS were defined as patients whom the procedures were performed on; RNs were the individuals performing the procedures.
  Hospital Standard of Care: Standard of Care for PIVC access per hospital protocol
- Stage 2 Education: RN education and training in the use of B. Braun PIVC products, devices and procedures.
  B. Braun Peripheral Advantage (PA) Program: B. Braun PA includes: Christie VeinViewer® Vision2 , Introcan Safety® IV Catheters, STEADYCare™ Smallbore Extension Set, and the PA Education
  **THIS PHASE WAS NOT CONDUCTED**
- Stage 3 Run-In: Familiarization of study RNs with the B. Braun devices and procedures in a clinical setting.
  B. Braun Peripheral Advantage (PA) Program: B. Braun PA includes: Christie VeinViewer® Vision2 , Introcan Safety® IV Catheters, STEADYCare™ Smallbore Extension Set, and the PA Education
  **THIS PHASE WAS NOT CONDUCTED**
- Stage 4 Post-Education: Study site uses B. Braun PIVC device(s) and procedure(s) on patients.
  B. Braun Peripheral Advantage (PA) Program: B. Braun PA includes: Christie VeinViewer® Vision2 , Introcan Safety® IV Catheters, STEADYCare™ Smallbore Extension Set, and the PA Education
  **THIS PHASE WAS NOT CONDUCTED**
Period: Overall Study
Arm/Group | Stage 1 Baseline | Stage 2 Education | Stage 3 Run-In | Stage 4 Post-Education
Started | 43 | 0 | 0 | 0
Completed | 43 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated during stage 1 for recruitment futility. Stages 2 through 4 were not conducted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Baseline | Stage 2 Education | Stage 3 Run-In | Stage 4 Post-Education | Total
Number analyzed (Participants) | 44 | 0 | 0 | 0 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (16.15) |  |  |  | 69.2 (16.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 |  |  |  | 27
  Male | 17 |  |  |  | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  | 0
  Not Hispanic or Latino | 44 |  |  |  | 44
  Unknown or Not Reported | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  | 0
  Asian | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
  Black or African American | 0 |  |  |  | 0
  White | 44 |  |  |  | 44
  More than one race | 0 |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 |  |  |  | 44
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (9.47) |  |  |  | 31.9 (9.47)

OUTCOME MEASURES:

1. Primary Outcome: Complications Associated With PIVC Use
Description: [Planned] Outcome: Evaluate the impact of B. Braun Peripheral Advantage (PA) Program on the number of stick attempts with complications associated with PIVC use.
  Due to the early termination in Stage 1, no data were collected from Stages 2 through 4 to perform comparative analyses.
Time Frame: Through study completion, an estimate of 1 year
Population: Study stopped due to recruitment futility. Stages 2 through 4 were not conducted.
Measure: Count of Units; unit: Stick Attempts
Units Other Than Participants: Stick Attempts
Arm/Group | Stage 1 Baseline | Stage 2 Education | Stage 3 Run-In | Stage 4 Post-Education
Number analyzed (Participants) | 43 | 0 | 0 | 0
Number analyzed (Stick Attempts) | 57 | 0 | 0 | 0
Stick Attempts | 22 |  |  |

2. Secondary Outcome: Catheter Indwell Time
Description: Evaluate the effect of B. Braun PA on catheter indwell time associated with catheter insertion.
Time Frame: Up to 48 hours and between 48 and 168 hours
Population: Study stopped due to recruitment futility. Stages 2 through 4 were not conducted.
  Of the 43 patients with attempted needle sticks, only 35 were successful.
Measure: Median (Full Range); unit: Hours
Arm/Group | Stage 1 Baseline | Stage 2 Education | Stage 3 Run-In | Stage 4 Post-Education
Number analyzed (Participants) | 35 | 0 | 0 | 0
Hours
  < 48 hours | 25.00 [2.37 to 47.68] |  |  |
  >= 48 hours | 76.84 [48.42 to 211.35] |  |  |

3. Secondary Outcome: First Attempt Success Rates (First Stick Success)
Description: Evaluate the effect of B. Braun PA on first attempt success rates (first stick success) associated with catheter insertion.
Time Frame: Initial needle stick (baseline)
Population: Study stopped due to recruitment futility. Stages 2 through 4 were not conducted.
Measure: Count of Units; unit: Stick Attempts
Units Other Than Participants: Stick Attempts
Arm/Group | Stage 1 Baseline | Stage 2 Education | Stage 3 Run-In | Stage 4 Post-Education
Number analyzed (Participants) | 43 | 0 | 0 | 0
Number analyzed (Stick Attempts) | 57 | 0 | 0 | 0
Stick Attempts | 28 |  |  |

4. Secondary Outcome: Aggregate Costs Associated With Catheter Insertion
Description: Evaluate the effect of B. Braun PA on aggregate costs associated with catheter insertion.
Time Frame: Through study completion, an estimate of 1 year
Population: Data were not collected for this Outcome Measure as a consequence of not performing the assessment. Study stopped during Stage 1 due to recruitment futility.
Arm/Group | Stage 1 Baseline | Stage 2 Education | Stage 3 Run-In | Stage 4 Post-Education
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Each subject/patient was assessed from baseline (initial needle stick) up to 168 hours (longest catheter indwell time reported).
Description: Study stopped during Stage 1 due to recruitment futility. Stages 2 through 4 were not conducted.
Arm/Group | Stage 1 Baseline | Stage 2 Education | Stage 3 Run-In | Stage 4 Post-Education
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 12/43 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Baseline (N=43) | Stage 2 Education (N=0) | Stage 3 Run-In (N=0) | Stage 4 Post-Education (N=0)
Infiltration (General disorders) | 4 | 0 | 0 | 0
Occlusion (Product Issues) | 3 | 0 | 0 | 0
Accidental Removal (Surgical and medical procedures) | 4 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to limitations in the data collected only in Stage 1, no conclusions can be drawn on the impact of B. Braun PA Program on the incidence of complications associated with PIVC use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications and redact proprietary information prior to public release and can embargo communications regarding trial results for a period of at least 45 days from the time submitted to the sponsor for review. The sponsor cannot require changes (other than as described) to the communication however the embargo may be extended an additional 60 days if patent issues are involved.

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT04048863/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT04048863/SAP_001.pdf